CLINICAL TRIAL: NCT04477525
Title: The Feasibility of Performing Erector Spinae (ESP) Nerve Block in Bariatric Patients; a Case Series Stud
Brief Title: The Feasibility of Performing Erector Spinae (ESP) Nerve Block in Bariatric Patients; a Case Series Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI changed hospital center
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11082
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Nerve Pain
MeSH Terms: conditions — Neuralgia | interventions — Parapsychology; Nerve Block; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP nerve block (Experimental)
  Interventions: Procedure: Ultrasound Guided Erector Spinae Plane (ESP) Nerve Block; Drug: Bupivacaine Injection
- Standard of Care (No Intervention): Standard of care includes IV opioids, NSAIDs (commonly ketorolac), +/- acetaminophen. No regional anesthesia will be given to control patients.

INTERVENTIONS:
Procedure: Ultrasound Guided Erector Spinae Plane (ESP) Nerve Block — The planned intervention is a bilateral erector spinae nerve block for patients undergoing bariatric surgery. This intervention will be performed in the PACU for patients with an NRS pain score >5. All eligible candidates who have consented for this study will be present in the PACU, have all standard ASA monitoring placed. The patient will then be placed in a sitting position. The patient will then be prepped with chlorhexidine in the thoracic region and draped in a sterile fashion. The ultrasound will be brought in over the patient and the T7 Transverse Processes (TP) will be identified. An echogenic needle will be placed under direct ultrasound guidance on the TP. Then, 20 cc of 0.25% bupivacaine will be injected.
  Arms: ESP nerve block
Drug: Bupivacaine Injection — 20 cc of 0.25% bupivacaine will be injected
  Arms: ESP nerve block

SUMMARY:
This study is a pilot study to assess the effectiveness of erector spinae (ESP) nerve blocks for postoperative pain control following bariatric surgery. Currently, there are mainly case series/pilot studies describing the use of ESP nerve blocks for postoperative pain control in abdominal procedures; of these only one uses this treatment modality for bariatric procedures. The population undergoing bariatric surgery poses specific challenges to postoperative pain management. They often have comorbid obstructive sleep apnea, which puts them at greater risk for ventilatory depression when treated with parenteral opioids. This risk can be reduced with regional techniques. The ESP nerve blocks provide visceral and somatic pain coverage as opposed to the more commonplace transversus abdominis plane nerve block which only provides somatic coverage. This means that the ESP nerve blocks will cover incisional pain as well as the discomfort associated with the pain from the procedure itself. This study intends to build on current knowledge by proving that the use of ESP in the post-operative are providing a significant reduction in pain scores as well as reducing the need for parenteral opioids. Thus, decreasing the risk of postoperative ventilatory complications.

In preparation for this study, three pilot studies were reviewed. The studies assessed the usefulness of ESP nerve blocks on patients undergoing abdominal surgery. Single-shot bilateral ESP blocks were performed in the first two studies. One of the studies, patients undergoing ventral hernia repair and the other for patients undergoing bariatric surgery. The third pilot study used bilateral ESP blocks followed by a continuous infusion on one patient undergoing an open prostatectomy with bladder reconstruction. All the ESP blocks were placed preoperatively at the T7 transverse process. In the studies using a single shot technique 20-30 ml of ropivacaine 0.5% was used. For the continuous ESP catheter an initial bolus of bupivacaine 0.25% 10 mls followed by continuous infusion rate of 6 ml/hr bilaterally. All showed a significant reduction numerical rating scale (NRS) as a primary outcome. The secondary outcome of reduced 24-hour parenteral opioid consumption was also achieved by all three studies.

ELIGIBILITY:
Inclusion Criteria:

* Age range 21 - 70.
* ASA II: A patient with mild systemic disease-ASA III: A patient with severe systemic disease
* Patients included are those immediately postoperative from bariatric surgery who have an NSR pain score >5

Exclusion Criteria:

* Patients excluded are those who are ASA IV or greater, refuse nerve block intervention,
* Diagnosis of any coagulopathy disorder,
* Allergy to local anesthetics,
* Have active infection over proposed injection sites.
* Patients with ASA >III was excluded due to overall health concerns of poorly controlled chronic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-22 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Rate of reduction of opiod usage after ESP Block | 24 hours
  This study will evaluate the role of ESP blocks in reducing 24-hour opioid requirements after bariatric surgery, specifically looking into 30% or more reduction in opioid usage ( morphine equivalence) in the 24 hours.

SECONDARY OUTCOMES:
Number of patients who experience an adverse events | Up to 3 days
Pain scores (self reported) assessed by the NRS rating scale | Every 30 min while in the post-anesthesia care unit (PACU); at 24 and 48 hours during hospital stay
  Pain scores will be collected every 30 mins in the PACU and at 24 and 48 hours during the hospital stay. NRS pain scale=0 no pain to 10 Worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Farah Fadi, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No